CLINICAL TRIAL: NCT05784831
Title: Development and Feasibility Test of an Ecological Momentary Intervention (EMI) - ReApp, to Promote and Improve Stress Resilience, Specifically to Increase Reappraisal.
Brief Title: Development and Feasibility Test of an Ecological Momentary Intervention (EMI) - ReApp, to Increase Reappraisal.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Radboud University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UZH_ReApp
Record Dates: First submitted 2022-05-25; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Stress
Keywords: stress; health; resilience

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Intervention Group (Experimental): Group using the app delivering reappraisal training for 21 consecutive days.
  Interventions: Device: Reappraisal training
- Burst Intervention Group (Experimental): Group using the app delivering reappraisal training for 7 consecutive days, then having 7 days break and again using the app 7 consecutive days.
  Interventions: Device: Reappraisal training
- Active Control Group (Active Comparator): Group using the ecological momentary assessment app for 21 consecutive days.
  Interventions: Device: Ecological Momentary Assessment

INTERVENTIONS:
Device: Reappraisal training — The EMI developed and tested here is based on theoretical and empirical findings and consists of several items and repeated training using various individual scenarios from participants' life that will be presented to participants via an app on their smartphones.
  Other Names: ReApp
  Arms: Burst Intervention Group; Regular Intervention Group
Device: Ecological Momentary Assessment — The EMA tested here collects data on participants' mood and behavior.
  Other Names: EMA
  Arms: Active Control Group

SUMMARY:
The aim of the current project is to develop and test Ecological Momentary Interventions (EMIs) to promote and improve stress resilience, specifically, an EMI to increase positive reappraisal.

EMIs are mostly smartphone-based applications that deliver interventions to people as they go about in their daily lives. The EMI tested here is based on theoretical and empirical findings and consists of several items and repeated training using various individual scenarios from participants' life that will be presented to participants via an app on their smartphones.

This study tests the efficacy of the EMI on a change in (i) reappraisal and (ii) indices of perceived stress. One hundred twenty healthy student participants, aged 18-29 will be invited to the study. Participants will be screened and those who score below 13 points of reappraisal skills in a Cognitive Emotion Regulation Questionnaire, will be included in the study. This is necessary in order to avoid a ceiling effect on reappraisal skills, which may be high in students.

Then, the participants will be randomly assigned to experimental (reappraisal EMI in regular and burst design) and control conditions (control EMA) and fill in questionnaires. The reappraisal EMI groups will be taught reappraisal skills and will be asked to apply them to personal situations repeatedly. The control EMA group will have the same app consisting of Ecological Momentary Assessment only. The training will last 21 consecutive days and the app will send (i) 5 prompts per day to ask about the current mood of the user in control and both experimental groups and (ii) at least two prompts per day resulting in a total of min. 42 reappraisal training sessions in the regular experimental group or 28 reappraisal training sessions in the burst experimental group. What is more, every participant has the possibility to trigger the EMA or EMI anytime they wish to. After using the app, participants will fill in some questionnaires again. The whole study will be conducted remotely (Video calls and app use) to avoid unnecessary COVID-related risks for participants.

ELIGIBILITY:
Inclusion Criteria:

1. being a student
2. having sufficient knowledge of the German language
3. being a smartphone user
4. low results in a CERQ questionnaire (less than 13 points in the Positive Reappraisal subscale).

Exclusion Criteria:

(1) having a current mental illness reported in the screening process.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | 21 days
  Self-reported level of stress, scale range [0-40], higher score = worse outcome
Beck Depression Inventory II (BDI-II) | 21 days
  Self-reported depressive symptoms, scale range [0-63], higher score = worse outcome
Cognitive Emotion Regulation Questionnaire (CERQ) | 21 days
  Self-reported reappraisal skills, scale range [5-20], higher score = better outcome
State-Trait Anxiety Inventory (STAI) | 21 days
  Self-reported anxiety symptoms, scale range [20-80], higher score = worse outcome
Emotion Regulation Questionnaire (ERQ) | 21 days
  Self-reported reappraisal use, scale range [6-42], higher score = better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Kleim, PhD, Principal Investigator — University of Zurich
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
OSF
Supporting Information: CSR
Time Frame: from August 2022 onwards
Access Criteria: open to everyone